CLINICAL TRIAL: NCT04059185
Title: Longitudinal Follow-up of Brief Parenting Interventions to Reduce Risk of Child Physical Maltreatment in a Selected Population
Brief Title: Longitudinal Follow-up of Brief Parenting Interventions to Reduce Risk of Child Physical Maltreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Vanderbilt University Medical Center (Other); Boston College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 492966; R01HD093665 (NIH)
Record Dates: First submitted 2019-07-31; First posted 2019-08-16 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-09

CONDITIONS: Parenting; Child Behavior; Child Rearing
Keywords: Child abuse; Child maltreatment
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Program 1 (Experimental): Triple P-Level 2 (TPL2), parenting education and consultation
  Interventions: Other: Triple P-Level 2
- Program 2 (Experimental): Play Nicely (PN), multimedia, computer-based parenting education
  Interventions: Other: Play Nicely
- Control (Placebo Comparator): Our "usual care" control group participants receive a resource and referral list for local social services
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Triple P-Level 2 — Triple P-Level 2 (TPL2) consists of a brief, 30 minute, one-on-one consultation with a parenting professional followed by a phone call from that professional roughly 2 weeks later. TPL2 will be delivered on an individual level and consist of a brief, 20 to 40 minute, one-on-one parenting consultation. Parents will receive a positive parenting booklet. They also will be offered parenting tip sheets that are designed to provide basic information on the prevention and management of common behavioral, emotional and developmental problems. All materials are: 1) written in simple English; 2) understandable at a sixth grade reading level; 3) gender-sensitive; and 4) avoid technical and colloquial expression that may pose barriers from non-English speaking backgrounds. Participants will receive a follow-up phone call to check on the family's progress and offer any additional needed advice.
  Arms: Program 1
Other: Play Nicely — Play Nicely is a brief, multimedia, computer-based educational program. The online program uses narrated modules to enhance parenting skills and promote effective parental responses to normal aggressive behavior in young children. The parent educational module presents a hypothetical situation of one child harming another. As the module progresses the viewer is given 20 different discipline options from which to choose. Participants are encouraged to click on all the options they wish to learn more about. The different options provide ways to respond to the situation and explain that there are discipline choices that are considered "Great options," "Good options after others have been tried," or "There are better options." The length of the program is dependent on how many of the 20 discipline options the participant chooses to learn about, but generally it can be finished in 20-40 minutes.
  Arms: Program 2
Other: Usual care — Our "usual care" control group participants receive a resource and referral list for local social services
  Arms: Control

SUMMARY:
Universal and broad selective parenting education programs that improve parenting skills, increase parents' understanding of child development, and teach positive child discipline strategies can prevent use of corporal punishment and child physical maltreatment. The proposed research addresses this critical need by investigating brief, relatively low-resource intensive primary prevention parenting programs that can be disseminated widely. By reducing cumulative adverse childhood experiences, which include child physical maltreatment, these interventions are expected to reduce long-term health disparities and risks for major public health problems, such as violence, smoking, obesity, drug abuse, risky sexual behavior, mental health disorders, and heart disease, among others

DETAILED DESCRIPTION:
1. Study design

   Our long-term goal is to enlarge the evidence base for low resource-intensive and widely adaptable interventions that effectively target parenting outcomes to reduce risk of child physical abuse in settings with broad reach. The objective of this study is to test the effectiveness of two such interventions in promoting effective parenting and reducing child physical abuse risk as compared with "usual care" parenting education. The central hypothesis is that each of two brief interventions, Triple P-L2 and Play Nicely, will be more effective in improving parenting effectiveness and reducing child behavioral and emotional problems than the "usual care" condition. Full scale Triple-P is an evidence-based, five-level system of interventions shown to reduce risk for child maltreatment when all 5 levels are implemented. However, implementation of a single level would be much less costly, more easily disseminated, and might in itself reduce risk in a broader population. Play Nicely is a brief computer-based intervention that has shown preliminary evidence for shifting attitudes about use of physical discipline when implemented in a pediatric primary care setting. However, it has yet to be tested within a large randomized-controlled trial (RCT). The rationale for this study is to be able to inform policy for parent service or clinic centers serving high-volumes of parents that are interested in adopting relatively low-resource intensive interventions in order to reduce risk of child physical abuse and improve child health and development trajectories.

   This is a community-based RCT. Parents (n=1200) with children 2 to 7 years of age will be recruited from local Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) clinics and by open recruitment. Once consented, they will be enrolled, a baseline interview will be conducted, and they will be randomly assigned to one of 3 conditions: (1) Triple P-Level 2 only (L2) intervention, (2) Play Nicely intervention, or (3) a "usual care" control group. Three months later, a follow-up interview will be conducted in order to test for intervention effects. In addition, a long term follow-up will be conducted to test sustained effects of the intervention. Participants' children (n=1200) will be enrolled for the long term follow-up. Children will be invited to participate in order for the adult participant to be observed interacting with the child in several very benign behavioral activities. Adult participants that do not want to enroll their child may participate in the long term follow-up survey which they will have previously consented to. Our study name for presentation in the local community is "Tulane Innovations in Positive Parenting Study" (TIPPS).
2. Subject Population

   We will recruit a total number of 2400 participants for this study. We will recruit 1200 adult participants from City of New Orleans and Jefferson Parish WIC Clinics. During the long-term follow-up visit, one child for each adult with be enrolled (n=1200).
3. Procedure

Recruitment: Recruitment has taken place in WIC clinic waiting rooms. If a parent is eligible and interested, the TIPPS Staff Member will then confirm that she has completed all necessary WIC documentation and that she is scheduled for a follow-up appointment with WIC before moving forward with consent and enrollment.

Baseline Interview: After the participant is taken through the informed consent process, a TIPPS Team Member will then conduct the Baseline interview. Once the Baseline Interview is complete (approximately 45 minutes), the participant will be informed of their random assignment to one of three conditions: (1) Triple P-Level 2, (2) Play Nicely, or (3) Control. The next procedure will then depend upon which of the three groups the person is assigned to. (See "Arms and Interventions" section for more details.) Debrief: Once both the Baseline Interview and the Intervention phase are complete, a TIPPS Team Member will schedule the 3-month Follow-Up Appointment, provide the control condition, provide an area-specific resource guide, and give the participant our incentive. The whole procedure (enrollment, baseline interview, intervention, and debrief) is expected to take no more than 2 hours.

3-Month Follow-Up Visit: If the participant has a WIC appointment, when they return to WIC for their 3-month visit and once they've completed their WIC documentation, a TIPPS Team Member will conduct the 3-month interview with them. This interview should take no more than 45 minutes. As with the baseline visit, childcare will be offered when available and the Suicide Risk Protocol will be followed if needed. In the event that the participant cannot return to the study site for their 3-month visit, the TIPPS team member will schedule the 3-Month interview as a phone interview. If the participant is unwilling or unable to complete the follow-up interview over the phone, a follow-up interview will be scheduled at a more convenient location for the participant, such as a local business or the participant's home.

The long term follow-up visit protocol described below is possible due to funding from NICHD which will fund this study from 7/2018 - 6/2023.

Long Term Follow-Up Visit : Participants will be asked to arrive at the research site with their child indicated as the index child in the baseline survey visit. A trained research team member will conduct the informed consent procedures followed at the baseline visit. If the adult participate does not want her child to participate, she may complete the long-term follow-up survey which she has consented to previously. If she agrees to participate and gives permission for her child to participate, she must review and sign a new consent form before participating in any Long Term Follow-Up activities. The informed consent form will be a record of the mother's agreement for both her and her child to participate. Upon completion of the informed consent process, a research assistant will conduct the Long Term Follow-Up interview with the adult participant. A separate research assistant will engage the child participant in several tasks. The first task will be the NIH Toolbox, which measures Cognitive flexibility and executive function, administered by tablet. Next, the child will be given the Marshmallow Test, which is an inhibitory control task where the child is told to wait for to eat a marshmallow until the research assistant returns to the room, and if they are able to wait, they will get two marshmallows. The time before the child eats the marshmallow is a validated measure of inhibitory control; inhibitory control has been found to be a significant predictor of child health and development outcomes across the life course.

Following the surveys, ECG data will be collected on the child and mother concurrently, acquired using Mindware Technologies mobile recorders, and transmitted via wireless signals to a computer monitored by a research assistant. After participant and child leads have been connected to ECG machines, the participant and child will do 3 very benign behavioral activities together: 1) watch a short video, 2) tell a story together, and 3) engage in a cooperative task (drawing with an Etch A Sketch). Interactions will be video recorded with parental consent and child assent and coding of parent and child behaviors will be done using the coding interactive behavior (CIB) coding system. Respiratory Sinus Arrhythmia (RSA) values will be processed in 30-second epochs across tasks for mothers and for children, and multilevel growth models will be built examining each 30-second epoch over the course of the task, relative to the individuals' baseline RSA. Dr. Drury will have full oversight of the dyadic coding of video recorded interactions between mother and child. Lastly, a TIPPS Team Member will provide the participant with locally-based health care resources guide.

4. Benefits

There will be no direct benefits to subjects for participating in this research, but the knowledge gained from the study may benefit society in general. Anticipated benefits might include a participant's greater understanding of positive parenting techniques.

5. Costs

There will be no costs to the subject for participating in this research study.

6. Alternatives

Subjects always have the option to not participate in the research.

ELIGIBILITY:
Inclusion Criteria:

Adult participants must be:

* Women
* English-speaking
* adults, age 18 or older
* a parent of at least one child between 2 and 7 years of age
* a primary caregiver of that child
* able to return to WIC (or recruitment site) for follow-up 3 months later
* available for up to 2 hours on date of recruitment to complete the baseline visit

Child participants:

* must be the "index child" of the adult participant as indicated in the baseline interview
* all genders eligible

Exclusion Criteria:

* anyone who does not meet the above inclusion criteria

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1133 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Taylor, PhD, Principal Investigator — Boston College School of Social Work; Julia M Fleckman, PhD, Principal Investigator — Tulane University
Locations (1):
- Tulane University School of Public Health and Tropical Medicine, New Orleans, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Program 1 (Triple P-Level 2): Triple P-Level 2 (TPL2), parenting education and consultation
  Triple P-Level 2 (TPL2) consists of a brief, 30 minute, one-on-one consultation with a parenting professional followed by a phone call from that professional roughly 2 weeks later. TPL2 will be delivered on an individual level and consist of a brief, 20 to 40 minute, one-on-one parenting consultation. Parents will receive a positive parenting booklet. They also will be offered parenting tip sheets that are designed to provide basic information on the prevention and management of common behavioral, emotional and developmental problems. All materials are: 1) written in simple English; 2) understandable at a sixth grade reading level; 3) gender-sensitive; and 4) avoid technical and colloquial expression that may pose barriers from non-English speaking backgrounds. Participants will receive a follow-up phone call to check on the family's progress and offer any additional needed advice.
- Program 2 (Play Nicely): Play Nicely (PN), multimedia, computer-based parenting education
  Play Nicely is a brief, multimedia, computer-based educational program. The online program uses narrated modules to enhance parenting skills and promote effective parental responses to normal aggressive behavior in young children. The parent educational module presents a hypothetical situation of one child harming another. As the module progresses the viewer is given 20 different discipline options from which to choose. Participants are encouraged to click on all the options they wish to learn more about. The different options provide ways to respond to the situation and explain that there are discipline choices that are considered "Great options," "Good options after others have been tried," or "There are better options." The length of the program is dependent on how many of the 20 discipline options the participant chooses to learn about, but generally it can be finished in 20-40 minutes.
Period: Longitudinal Assessment-Adults Only
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Started | 289 | 294 | 297
Completed Baseline Survey and Study Condition | 272 | 271 | 280
Completed 3 Month Post-intervention Survey | 243 | 239 | 258
Completed 4 Year Post-intervention Survey | 142 | 133 | 165
Completed (This is the number of adults who completed all longitudinal assessments (4 year post-intervention clinic visit, 4 year post-intervention survey, 3 month post-intervention survey, and baseline); only 2 persons in this group did not complete the 3 month post-intervention survey) | 81 | 72 | 100
Not Completed | 208 | 222 | 197
Not completed — Lost to Follow-up | 187 | 195 | 177
Not completed — Protocol Violation | 11 | 13 | 13
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Baseline survey incomplete | 4 | 8 | 3
Not completed — Death | 4 | 4 | 3
Period: 4 Year Post-Intervention Clinic-Children
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Started (These numbers reflect the index children who were eligible to participate in the 4 year post-intervention clinic visit with their adult caregiver. Only those children whose adult caregiver agreed to partcipate in the 4 year post-intervention clinic visit were eligible.) | 81 | 72 | 100
Completed | 81 | 72 | 100
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Program 1 (Triple P-Level 2): Triple P-Level 2 (TPL2), parenting education and consultation
  Triple P-Level 2: Triple P-Level 2 (TPL2) consists of a brief, 30 minute, one-on-one consultation with a parenting professional followed by a phone call from that professional roughly 2 weeks later. TPL2 will be delivered on an individual level and consist of a brief, 20 to 40 minute, one-on-one parenting consultation. Parents will receive a positive parenting booklet. They also will be offered parenting tip sheets that are designed to provide basic information on the prevention and management of common behavioral, emotional and developmental problems. All materials are: 1) written in simple English; 2) understandable at a sixth grade reading level; 3) gender-sensitive; and 4) avoid technical and colloquial expression that may pose barriers from non-English speaking backgrounds. Participants will receive a follow-up phone call to check on the family's progress and offer any additional needed advice.
- Program 2 (Play Nicely): Play Nicely (PN), multimedia, computer-based parenting education
  Play Nicely: Play Nicely is a brief, multimedia, computer-based educational program. The online program uses narrated modules to enhance parenting skills and promote effective parental responses to normal aggressive behavior in young children. The parent educational module presents a hypothetical situation of one child harming another. As the module progresses the viewer is given 20 different discipline options from which to choose. Participants are encouraged to click on all the options they wish to learn more about. The different options provide ways to respond to the situation and explain that there are discipline choices that are considered "Great options," "Good options after others have been tried," or "There are better options." The length of the program is dependent on how many of the 20 discipline options the participant chooses to learn about, but generally it can be finished in 20-40 minutes.
- Total: Total of all reporting groups
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control | Total
Number analyzed (Participants) | 353 | 343 | 380 | 1076
Age, Categorical [Count of Participants; unit: Participants] — Population: The numbers entered for "adults" reflect the number of participants who completed the baseline portion of the overall study. The numbers of "index children" entered reflect those who participated in the 4 year post-intervention clinic visit (also known as the "dyadic visit").
  Participants
    Adults: number analyzed (Participants) | 272 | 271 | 280 | 823
    Adults: <=18 years | 1 | 0 | 0 | 1
    Adults: Between 18 and 65 years | 269 | 269 | 279 | 817
    Adults: >=65 years | 2 | 2 | 1 | 5
    Index children: number analyzed (Participants) | 81 | 72 | 100 | 253
    Index children: <=18 years | 81 | 72 | 100 | 253
    Index children: Between 18 and 65 years | 0 | 0 | 0 | 0
    Index children: >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The numbers entered for "adults" reflect the number of participants who completed the baseline portion of the overall study. The numbers of "index children" entered reflect those who participated in the 4 year post-intervention clinic visit (also known as the "dyadic visit").
  Participants
    Adults: number analyzed (Participants) | 272 | 271 | 280 | 823
    Adults: Female | 272 | 271 | 280 | 823
    Adults: Male | 0 | 0 | 0 | 0
    Index children: number analyzed (Participants) | 81 | 72 | 100 | 253
    Index children: Female | 39 | 40 | 54 | 133
    Index children: Male | 42 | 32 | 46 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The numbers entered for "adults" reflect the number of participants who completed the baseline portion of the overall study. The numbers of "index children" entered reflect those who participated in the 4 year post-intervention clinic visit (also known as the "dyadic visit").
  Participants
    Adults: number analyzed (Participants) | 272 | 271 | 280 | 823
    Adults: Hispanic or Latino | 18 | 19 | 19 | 56
    Adults: Not Hispanic or Latino | 194 | 197 | 195 | 586
    Adults: Unknown or Not Reported | 60 | 55 | 66 | 181
    Index children: number analyzed (Participants) | 81 | 72 | 100 | 253
    Index children: Hispanic or Latino | 0 | 0 | 0 | 0
    Index children: Not Hispanic or Latino | 0 | 0 | 0 | 0
    Index children: Unknown or Not Reported | 81 | 72 | 100 | 253
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The numbers entered for "adults" reflect the number of participants who completed the baseline portion of the overall study. The numbers of "index children" entered reflect those who participated in the 4 year post-intervention clinic visit (also known as the "dyadic visit").
  Participants
    Adults: number analyzed (Participants) | 272 | 271 | 280 | 823
    Adults: American Indian or Alaska Native | 1 | 0 | 0 | 1
    Adults: Asian | 3 | 1 | 3 | 7
    Adults: Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
    Adults: Black or African American | 231 | 232 | 239 | 702
    Adults: White | 16 | 13 | 16 | 45
    Adults: More than one race | 13 | 12 | 9 | 34
    Adults: Unknown or Not Reported | 7 | 13 | 13 | 33
    Index children: number analyzed (Participants) | 81 | 72 | 100 | 253
    Index children: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Index children: Asian | 0 | 0 | 0 | 0
    Index children: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Index children: Black or African American | 0 | 0 | 0 | 0
    Index children: White | 0 | 0 | 0 | 0
    Index children: More than one race | 0 | 0 | 0 | 0
    Index children: Unknown or Not Reported | 81 | 72 | 100 | 253
Region of Enrollment [Number; unit: participants] — Population: The numbers entered reflect the overall study. All participants, including the index children who comprise part of the sample at the 4 year post-intervention clinic visit, all resided in the same region, the United States.
  participants
    United States | 353 | 343 | 380 | 1076

OUTCOME MEASURES:

1. Primary Outcome: Parent - Change From Baseline Frequency of Corporal Punishment Use at 3 Months and at Long-term Follow-up
Description: The measure was collected at baseline, 3 month post-intervention, and 4 year post-intervention. This question asks participants "How often on average in the past month have you spanked your child?" with seven categories: 0) never, 1) once or twice in the past month, 2) about once a week, 3) about twice a week, 4) about once every other day, 5) about once a day, and 6) more than once a day. Using the 0-6 score response range, the outcome was calculated by subtracting the baseline score from the 3 month or 4 year post-intervention score, such that a negative score indicates decrease in frequency of spanking at the post-intervention timepoint.
Time Frame: Baseline, 3 months post-intervention, 4 years post-intervention
Population: All available survey data for each time point was used. The baseline to 4 year post-intervention "number analyzed" differs from the baseline to 3 month post-intervention due to study attrition (lost to follow-up).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 242 | 239 | 258
score on a scale
  Baseline to 3 month post-intervention | -.32 (1.6) | -.27 (1.4) | -.17 (1.4)
  Baseline to 4 years post-intervention: number analyzed (Participants) | 143 | 134 | 166
  Baseline to 4 years post-intervention | -.69 (1.5) | -.68 (1.6) | -.80 (1.8)

2. Primary Outcome: Parent - Change From Baseline Attitudes Toward Use of Corporal Punishment at 3 Months and at Long-term Follow-up
Description: The Attitudes Towards Spanking (ATS) scale was collected at baseline, 3 months post-intervention, and 4 years post-intervention. The scale score response range was 0-28, with a higher number being stronger support for spanking. This change outcome was calculated by subtracting the baseline score from the 3 month or 4 year post-intervention score, such that a negative score indicates a decrease in approval of spanking at the post-intervention time point.
Time Frame: Baseline, 3 months post-intervention, 4 years post-intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 241 | 237 | 253
score on a scale
  Baseline to 3 month post-intervention | -.86 (5.8) | -2.1 (6.0) | -.13 (5.0)
  Baseline to 4 years post-intervention: number analyzed (Participants) | 142 | 132 | 162
  Baseline to 4 years post-intervention | -1.8 (6.6) | -2.5 (7.1) | -1.9 (6.3)

3. Secondary Outcome: Parent - Child Discipline Practices
Description: The Parental Discipline scale of the Parenting and Family Adjustment Scale (PAFAS) was collected at baseline, 3 month follow up, and long-term follow-up. This scale ranges from 0-54, with a higher number indicating more positive parenting.
Time Frame: Baseline, 3 months post-intervention, 4 years post-intervention
Population: All available survey data for each time point was used. The baseline, 3 month post-intervention, and 4 year post-intervention "number analyzed" differs due to study attrition (lost to follow-up).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 268 | 271 | 280
score on a scale
  Baseline | 44.1 (4.9) | 44.1 (4.8) | 45 (4.6)
  3 month post-intervention: number analyzed (Participants) | 241 | 236 | 258
  3 month post-intervention | 45.1 (5.3) | 44.9 (5.1) | 44.7 (4.9)
  4 years post-intervention: number analyzed (Participants) | 143 | 132 | 166
  4 years post-intervention | 43.7 (5.8) | 44.2 (5.7) | 44.5 (5.3)

4. Secondary Outcome: Child - Behavioral and Emotional Adjustment
Description: The Child Adjustment and Parent Efficacy Scale (CAPES) scale was collected at baseline, 3 month follow-up, and long-term follow-up. This scale ranges from 0-81, with a higher number indicating increased levels of emotional or behavioral problems.
Time Frame: Baseline, 3 months post-intervention, 4 years post-intervention
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 268 | 267 | 279
score on a scale
  Baseline | 21 (12.3) | 21.5 (12.5) | 20.8 (12.8)
  3 month post-intervention: number analyzed (Participants) | 240 | 238 | 256
  3 month post-intervention | 18.9 (11.9) | 20.6 (11.8) | 20.6 (12.6)
  4 years post-intervention: number analyzed (Participants) | 141 | 134 | 166
  4 years post-intervention | 17.2 (12) | 19.3 (13.8) | 17.9 (14.5)

5. Secondary Outcome: Child - Externalizing, Internalizing, and Total Symptoms
Description: The 113 item Child Behavior Checklist (CBCL) scale was collected at 4 year long-term follow-up. The outcome is a T-score calculated for total symptoms, with a higher score indicating more internalizing and externalizing behaviors. For the T-score of the CBCL, the population mean is 50 and the standard deviation is 10. T-Scores less than 60 are considered to be in the normal range, the borderline range consists of T-scores of 60-63, and the clinical range consists of T-scores greater than 63.
Time Frame: 4 years post-intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 137 | 126 | 162
T-score | 51.1 (11) | 51.2 (10.9) | 51.3 (13.3)

6. Secondary Outcome: Parent Sensitivity
Description: The outcome measure reported is the parent sensitivity score of the Coding Interactive Behavior (CIB) global rating scheme, during a challenge task and a social interaction task. Scores have a possible range of 1-115. A higher score indicates a higher level of parent sensitivity from caregiver to child.
Time Frame: 4 years post-intervention
Population: These numbers reflect the 236 adult participants within the adult-child dyads (n=236 total dyads) that completed the 4-year post-intervention clinic visit. No data is available for adult participants from 17 of the adult-child dyads because they did not consent to videotaped observation (n=11) or their data was invalid based on coding specifications (N=6).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 75 | 68 | 93
score on a scale
  Challenge task at the 4 years post-intervention clinic visit | 67.34 (14.82) | 68.43 (14.23) | 69.03 (14.49)
  Social interaction task at the 4 years post-intervention clinic visit | 72.75 (15.48) | 73.15 (15.63) | 70.68 (18.50)

7. Secondary Outcome: Child Social Involvement
Description: The outcome measure reported is the child social involvement score of the Coding Interactive Behavior (CIB) global rating scheme, during a challenge task and a social interaction task. Scores have a possible range of 1-70. A higher score indicates a higher level of child social involvement from caregiver to child.
Time Frame: 4 years post-intervention
Population: These numbers reflect the child participants within the adult-child dyads (n=236 total dyads) that completed the 4-year post-intervention clinic visit. No data is available for child participants from 17 of the adult-child dyads because they did not consent to videotaped observation (n=11) or their data was invalid based on coding specifications (N=6).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 75 | 68 | 93
score on a scale
  Challenge task at the 4 years post-intervention clinic visit | 46.16 (6.66) | 47.39 (6.84) | 47.27 (6.23)
  Social interaction task at the 4 years post-intervention clinic visit | 48.91 (11.79) | 50.18 (11.54) | 50.24 (11.90)

8. Secondary Outcome: Child Negative Emotionality
Description: The outcome measure reported is the child negative emotionality score of the Coding Interactive Behavior (CIB) global rating scheme, during a challenge task and a social interaction task. Scores have a possible range of 1-30. A higher score indicates a higher level of child negative emotionality from child.
Time Frame: 4 years post-intervention
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 75 | 68 | 93
score on a scale
  Challenge task at the 4 years post-intervention clinic visit | 8.43 (2.44) | 8.01 (1.93) | 8.21 (2.04)
  Social interaction task at the 4 years post-intervention clinic visit | 10.13 (3.58) | 9.77 (3.18) | 9.76 (3.38)

9. Secondary Outcome: Dyadic Negative States
Description: The outcome measure reported is the dyadic negative states score of the Coding Interactive Behavior (CIB) global rating scheme, during a challenge task and a social interaction task. Scores have a possible range of 1-10. A higher score indicates a higher level of dyadic negative states between caregiver and child.
Time Frame: 4 years post-intervention
Population: These numbers are adult-child dyads (n=236 total dyads, adults [n=236], and index children [n=236]) that completed the 4-year post-intervention clinic visit. No data is available for 17 dyads because they did not consent to videotaped observation (n=11) or their data was invalid based on coding specifications (N=6).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 75 | 68 | 93
score on a scale
  Challenge task at the 4 years post-intervention clinic visit | 3.36 (1.61) | 3.16 (1.46) | 3.06 (1.52)
  Social interaction task at the 4 years post-intervention clinic visit | 3.41 (1.40) | 3.37 (1.54) | 3.58 (1.84)

10. Secondary Outcome: Dyadic Reciprocity
Description: The outcome measure reported is the dyadic reciprocity score of the Coding Interactive Behavior (CIB) global rating scheme, during a challenge task and a social interaction task. Scores have a possible range of 1-15. A higher score indicates a higher level of dyadic reciprocity between caregiver and child.
Time Frame: 4 years post-intervention
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 75 | 68 | 93
score on a scale
  Challenge task at the 4 years post-intervention clinic visit | 3.11 (1.09) | 3.41 (1.03) | 3.23 (.99)
  Social interaction task at the 4 years post-intervention clinic visit | 3.01 (.90) | 3 (.94) | 3.01 (1.05)

11. Secondary Outcome: Parent Limit Setting
Description: The outcome measure reported is the parent limit setting score of the Coding Interactive Behavior (CIB) global rating scheme, during a challenge task and a social interaction task. Scores have a possible range of 1-35. A higher score indicates a higher level of parent limit setting from caregiver.
Time Frame: 4 years post-intervention
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 75 | 68 | 93
score on a scale
  Challenge task at the 4 years post-intervention clinic visit | 29.72 (3.76) | 29.69 (4.27) | 30.11 (3.27)
  Social interaction task at the 4 years post-intervention clinic visit | 27.24 (4.78) | 27.86 (4.51) | 26.64 (5.53)

12. Secondary Outcome: Child Compliance
Description: The outcome measure reported is the child compliance score of the Coding Interactive Behavior (CIB) global rating scheme, during a challenge task and a social interaction task. Scores have a possible range of 1-20. A higher score indicates a higher level child compliance.
Time Frame: 4 years post-intervention
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 75 | 68 | 93
score on a scale
  Challenge task at the 4 years post-intervention clinic visit | 14.87 (2.57) | 15.35 (2.01) | 15.19 (2.05)
  Social interaction task at the 4 years post-intervention clinic visit | 13.85 (2.59) | 14.24 (2.61) | 14.27 (2.42)

13. Secondary Outcome: Parent Baseline RSA
Description: The outcome measure is the average respiratory sinus arrhythmia (RSA) during the baseline task for the caregiver. RSA is a biomarker that typically ranges from 1-10 depending on the participant's physiology, with a higher number indicating greater variability between interbeat intervals during the task.
Time Frame: 4 years post-intervention
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 72 | 66 | 92
ms^2 | 6.01 (1.48) | 5.85 (1.54) | 5.75 (1.37)

14. Secondary Outcome: Child Baseline RSA
Description: The outcome measure is the average respiratory sinus arrhythmia (RSA) during the baseline task for the child. RSA is a biomarker that typically ranges from 1-10 depending on the participant's physiology, with a higher number indicating greater variability between interbeat intervals during the task.
Time Frame: 4 years post-intervention
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 76 | 62 | 90
ms^2 | 7.01 (1.15) | 6.93 (1.11) | 7.00 (1.27)

15. Secondary Outcome: RSA Synchrony Challenge Task
Description: Respiratory sinus arrhythmia (RSA)
Time Frame: 4 years post-intervention
Reporting Status: Not Posted, anticipated posting 2025-06

16. Secondary Outcome: RSA Lead/Lag During Challenge Task
Description: Respiratory sinus arrhythmia (RSA)
Time Frame: 4 years post-intervention
Reporting Status: Not Posted, anticipated posting 2025-06

17. Secondary Outcome: Parent RSA During Challenge Task
Description: The outcome measure is the average respiratory sinus arrhythmia (RSA) during the challenge task for the caregiver. RSA is a biomarker that typically ranges from 1-10 depending on the participant's physiology, with a higher number indicating more variability in time between each heartbeat during the task.
Time Frame: 4 years post-intervention
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 71 | 65 | 91
ms^2 | 5.65 (1.36) | 5.47 (1.34) | 5.45 (1.30)

18. Secondary Outcome: Child RSA During Challenge Task
Description: The outcome measure is the average respiratory sinus arrhythmia (RSA) during the challenge task for the child. RSA is a biomarker that typically ranges from 1-10 depending on the participant's physiology, with a higher number indicating more variability in time between each heartbeat during the task.
Time Frame: 4 years post-intervention
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 77 | 62 | 92
ms^2 | 6.73 (1.14) | 6.72 (.99) | 6.63 (1.23)

19. Secondary Outcome: RSA Synchrony During Social Interaction Task
Description: Respiratory sinus arrhythmia (RSA)
Time Frame: 4 years post-intervention
Reporting Status: Not Posted, anticipated posting 2025-06

20. Secondary Outcome: RSA Lead/Lag During Social Interaction Task
Description: Respiratory sinus arrhythmia (RSA)
Time Frame: 4 years post-intervention
Reporting Status: Not Posted, anticipated posting 2025-06

21. Secondary Outcome: Parent RSA During Social Interaction Task
Description: The outcome measure is the average respiratory sinus arrhythmia (RSA) during the social interaction task for the caregiver. RSA is a biomarker that typically ranges from 1-10 depending on the participant's physiology, with a higher number indicating more variability in time between each heartbeat during the task.
Time Frame: 4 years post-intervention
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 72 | 64 | 91
ms^2 | 5.95 (1.31) | 5.76 (1.49) | 5.78 (1.25)

22. Secondary Outcome: Child RSA During Social Interaction Task
Description: The outcome measure is the average respiratory sinus arrhythmia (RSA) during the social interaction task for the child. RSA is a biomarker that typically ranges from 1-10 depending on the participant's physiology, with a higher number indicating more variability in time between each heartbeat during the task.
Time Frame: 4 years post-intervention
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 77 | 61 | 91
ms^2 | 6.76 (1.12) | 6.62 (1.11) | 6.71 (1.26)

23. Secondary Outcome: Child - Cognitive Flexibility
Description: The outcome measure is the age-corrected scale score of cognitive flexibility (Dimensional Change Card Sort) computed by the NIH Toolbox software. The score is standardized such that the mean score in the overall population is 100 and the standard deviation is 15, with scores above 100 being above the average performance for children of the indicated age.
Time Frame: 4 years post-intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 80 | 71 | 98
T-score | 89.9 (14.8) | 89.9 (14.2) | 88.8 (14.7)

24. Secondary Outcome: Child - Delay Time
Description: Behavioral inhibitory control/ marshmallow task
Time Frame: 4 years post-intervention
Population: This test is only valid for children that have not yet begun first grade. Due to a later than expected commencement of our data collection at the 4 year post-intervention clinic visit, none of the children in our study met this requirement and hence the test was not administered.
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 0 | 0 | 0

25. Secondary Outcome: Child - Executive Function
Description: The outcome measure is the age-corrected scale score of executive function (Flanker Inhibitory Control and Attention Test) computed by the NIH Toolbox software. The score is standardized such that the mean score in the overall population is 100 and the standard deviation is 15, with scores above 100 being above the average performance for children of the indicated age.
Time Frame: 4 years post-intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 80 | 70 | 99
T-score | 91.85 (16) | 85.8 (16.5) | 90.3 (14.1)

26. Secondary Outcome: Child - Distraction Strategy
Description: Behavioral inhibitory control/ marshmallow task
Time Frame: 4 years post-intervention
Population: as for outcome 24
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 0 | 0 | 0

27. Secondary Outcome: Child - Distress Level
Description: Behavioral inhibitory control/ marshmallow task
Time Frame: 4 years post-intervention
Population: as for outcome 24
Arm/Group | Program 1 (Triple P-Level 2) | Program 2 (Play Nicely) | Control
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the study period (from baseline through 4-year post-intervention).
Description: Adverse events and all-cause mortality are reported for all adult (n=880) and child participants (n=253).
Groups:
- Program 1 (Triple P-Level 2) - Adults: Triple P-Level 2 (TPL2), parenting education and consultation
  Triple P-Level 2: Triple P-Level 2 (TPL2) consists of a brief, 30 minute, one-on-one consultation with a parenting professional followed by a phone call from that professional roughly 2 weeks later. TPL2 will be delivered on an individual level and consist of a brief, 20 to 40 minute, one-on-one parenting consultation. Parents will receive a positive parenting booklet. They also will be offered parenting tip sheets that are designed to provide basic information on the prevention and management of common behavioral, emotional and developmental problems. All materials are: 1) written in simple English; 2) understandable at a sixth grade reading level; 3) gender-sensitive; and 4) avoid technical and colloquial expression that may pose barriers from non-English speaking backgrounds. Participants will receive a follow-up phone call to check on the family's progress and offer any additional needed advice.
- Program 2 (Play Nicely) - Adults: Play Nicely (PN), multimedia, computer-based parenting education
  Play Nicely: Play Nicely is a brief, multimedia, computer-based educational program. The online program uses narrated modules to enhance parenting skills and promote effective parental responses to normal aggressive behavior in young children. The parent educational module presents a hypothetical situation of one child harming another. As the module progresses the viewer is given 20 different discipline options from which to choose. Participants are encouraged to click on all the options they wish to learn more about. The different options provide ways to respond to the situation and explain that there are discipline choices that are considered "Great options," "Good options after others have been tried," or "There are better options." The length of the program is dependent on how many of the 20 discipline options the participant chooses to learn about, but generally it can be finished in 20-40 minutes.
- Control - Adults: Our "usual care" control group participants receive a resource and referral list for local social services
  Usual care: Our "usual care" control group participants receive a resource and referral list for local social services
- Program 1 (Triple P-Level 2) - Children: The index children of the parents who were assigned to Triple P-Level 2 (TPL2):
  Triple P-Level 2 (TPL2), parenting education and consultation
  Triple P-Level 2: Triple P-Level 2 (TPL2) consists of a brief, 30 minute, one-on-one consultation with a parenting professional followed by a phone call from that professional roughly 2 weeks later. TPL2 will be delivered on an individual level and consist of a brief, 20 to 40 minute, one-on-one parenting consultation. Parents will receive a positive parenting booklet. They also will be offered parenting tip sheets that are designed to provide basic information on the prevention and management of common behavioral, emotional and developmental problems. All materials are: 1) written in simple English; 2) understandable at a sixth grade reading level; 3) gender-sensitive; and 4) avoid technical and colloquial expression that may pose barriers from non-English speaking backgrounds. Participants will receive a follow-up phone call to check on the family's progress and offer any additional needed advice.
- Program 2 (Play Nicely) - Children: The index children of the parents who were assigned to Play Nicely (PN):
  Play Nicely: Play Nicely is a brief, multimedia, computer-based educational program. The online program uses narrated modules to enhance parenting skills and promote effective parental responses to normal aggressive behavior in young children. The parent educational module presents a hypothetical situation of one child harming another. As the module progresses the viewer is given 20 different discipline options from which to choose. Participants are encouraged to click on all the options they wish to learn more about. The different options provide ways to respond to the situation and explain that there are discipline choices that are considered "Great options," "Good options after others have been tried," or "There are better options." The length of the program is dependent on how many of the 20 discipline options the participant chooses to learn about, but generally it can be finished in 20-40 minutes.
- Control - Children: The index children of the parents who were assigned to control:
  Our "usual care" control group participants receive a resource and referral list for local social services
  Usual care: Our "usual care" control group participants receive a resource and referral list for local social services
Arm/Group | Program 1 (Triple P-Level 2) - Adults | Program 2 (Play Nicely) - Adults | Control - Adults | Program 1 (Triple P-Level 2) - Children | Program 2 (Play Nicely) - Children | Control - Children
All-Cause Mortality (participants affected / at risk) | 4/289 | 4/294 | 3/297 | 0/81 | 1/72 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/289 | 0/294 | 0/297 | 0/81 | 0/72 | 0/100
Other Adverse Events (participants affected / at risk) | 0/289 | 0/294 | 0/297 | 0/81 | 0/72 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT04059185/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT04059185/SAP_001.pdf